CLINICAL TRIAL: NCT02178423
Title: Ultrasound Guided Diagnosis of Central Venous Catheters in Children: A Feasibility Study
Brief Title: Feasibility Study of CVC Diagnosis Via Ultrasound in Children
Acronym: CVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Wolfgang Klug, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1059/2014; 1059/2014 (Other: Ethics committee Medical University of Vienna)
Record Dates: First submitted 2014-06-11; First posted 2014-06-30 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Ultrasound for Diagnosis of CVC Position in Children
Keywords: children, ultrasound, central catheter
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound (Experimental): Ultrasound for diagnosis of CVC position in children
  Interventions: Procedure: Ultrasound for diagnosis of CVC position in children

INTERVENTIONS:
Procedure: Ultrasound for diagnosis of CVC position in children — Using the ultrasound for diagnosis of the correct position of a central venous catheter in children immediate after the puncture.

SUMMARY:
After the placement of a central venous catheter in children, a routine chest X-ray will be performed in order to examine the correct position of the catheter. In this feasibility study the investigators intend to evaluate whether the ultrasound is as sufficient as the chest X-ray to verify the correct position of the central venous catheter in children with the purpose to prevent radiation on children in the future.

DETAILED DESCRIPTION:
For punctures of a central vein in very small children, ultrasound is an useful tool which allows for exact examination of the relevant anatomy in order to visualize the target vessel, so as to facilitate the puncture in real-time. However, to ascertain the correct position of the central venous catheter (CVC), a chest X-ray is still the gold standard. The main disadvantage of the X-ray is the children's exposure to radiation. That's why the investigators intend to perform this study whether the ultrasound is as sufficient as the chest X-ray to verify the correct position of a central venous catheter in children.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged between 0 and 8 years requiring a central venous catheter. The planned sample size is 20 subjects. The indication for a CVC, will be determined by the attending physician.

Inclusion criteria:

* Infants (inclusive early and late preterm) and children aged between 0 and 8 years
* Necessity of a central venous catheter
* Written informed consent given by parents after being provided with detailed information about the nature, risks, and scope of the catheterization
* No legal incapacity and/or other circumstances rendering the parents unable to understand the nature, scope and possible consequences of the catheterization

Exclusion Criteria:

* Parents refusal

Ages: 1 Day to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of the correct central venous catheter position. | After all patients have been included (three months), all clips of each participant will be presented to three blind observers, classifying these clips for two times and outcome measure will be assessed.
  Ultrasound imaging will be stored in mpeg format and deidentified for all examinations. The ultrasound movie will be split into five clips with a length of 5 seconds each (four clips with CVC not inserted but ultrasound head slightly moving and one clip with CVC in situ). The total of 110 clips is presented in random order to three blinded observers who classify these clips two times with a time gap of at least 2 weeks between the classifications.

SECONDARY OUTCOMES:
Exclusion of a pneumothorax via ultrasound compared to chest X-ray | At 30 to 60 minutes after central venous catheter insertion each participant will undergo chest ultrasound and chest X-ray.
  The chest X-ray and ultrasound will be performed in the post anesthesia care unit to rule out a pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Roth, Prof., Principal Investigator — Dep. of Anesthesia and Intensive Care Medicine
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria